CLINICAL TRIAL: NCT04147143
Title: Cabozantinib in Adult Patients With Advanced Renal Cell Carcinoma Following Prior Systemic Check Point Inhibition Therapy: a Retrospective, Non-interventional Study
Brief Title: CaboCHECK - Cabozantinib in Adult Patients With Advanced Renal Cell Carcinoma Following Prior Systemic Check Point Inhibition Therapy: a Retrospective, Non-interventional Study
Status: Terminated | Type: Observational
Why Stopped: Due to insufficient recruitment rate, recruitmend has been terminated after inclusion of 56 patients
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Other Study IDs: CaboCHECK
Record Dates: First submitted 2019-10-24; First posted 2019-10-31 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Advanced Renal Cell Carcinoma (All Subtypes); Metastatic Renal Cell Carcinoma (All Subtypes)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Documentation — Retrospective chart review of patients who have already completed treatment with cabozantinib after nivolumab or nivolumab plus ipilimumab before inclusion.

SUMMARY:
This is a non-interventional study to retrospectively evaluate the safety and to describe the effectiveness of cabozantinib after immunoncologic treatment with nivolumab or nivolumab plus ipilimumab in routine clinical practice. It consists of a retrospective chart review of patients who have already completed treatment with cabozantinib after nivolumab or nivolumab plus ipilimumab before inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject
2. Patients with advanced or metastatic renal cell carcinoma, including all subtypes
3. Age ≥ 18 years
4. Completion of treatment with nivolumab or nivolumab / ipilimumab combination therapy (any line of therapy) directly followed by cabozantinib treatment

Exclusion Criteria:

1. Patients who are unable to consent because they do not understand the nature, significance and implications of the observational trial
2. Involvement in the planning and / or conduct of the study (applies to both Ipsen staff and/or staff of sponsor and study site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥ 18 years with advanced or metastatic renal cell carcinoma (all subtypes) who have completed treatment with nivolumab or nivolumab plus ipilimumab (any line of systemic therapy) directly followed by cabozantinib treatment
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | through study completion, an average of 1 year
  Incidence of serious adverse events at least possibly related to cabozantinib treatment during and up to 30 days after the end of cabozantinib treatment

SECONDARY OUTCOMES:
number of dose reductions | through study completion, an average of 1 year
  number of dose reductions
number of dose interruptions | through study completion, an average of 1 year
  number of dose interruptions
number of terminations of cabozantinib treatment due to adverse events | through study completion, an average of 1 year
  number of terminations of cabozantinib treatment due to adverse events
ORR | through study completion, an average of 1 year
  ORR (investigator assessed; acc. RECIST v1.1 if available)
Clinical benefit rate (CBR) | through study completion, an average of 1 year
  Clinical benefit rate (CBR)
Duration of response | through study completion, an average of 1 year
  Duration of response in months
Duration of cabozantinib treatment | through study completion, an average of 1 year
  Duration of cabozantinib treatment in months
Time to next treatment | From date of last dose of cabozantinib until the date of first dose of next treatment, assessed up to 100 months
  Time to next treatment in months
Safety in IO-cabozantinib-sequence compared to cabozantinib single agent therapy historical data | through study completion, an average of 1 year
  Safety in IO-cabozantinib-sequence compared to cabozantinib single agent therapy historical data
Comparison of effectiveness endpoints of IO-cabozantinib-sequence to historical efficacy data (ORR, CBR) | through study completion, an average of 1 year
  Comparison of effectiveness endpoints of IO-cabozantinib-sequence to historical efficacy data (ORR, CBR)

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (2):
- Germany (2):
  - Uniklinik Essen, Essen, North Rhine-Westphalia
  - Uniklinik Münster, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared